CLINICAL TRIAL: NCT00002928
Title: A Phase II Trial of Paclitaxel Administered Weekly in Patients With Advanced Ovarian Cancer
Brief Title: Paclitaxel in Treating Patients With Recurrent or Progressive Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 96-070; CDR0000065361 (Registry Identifier: PDQ (Physician Data Query)); NCI-G97-1139
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients with recurrent or progressive advanced epithelial ovarian cancer following previous paclitaxel.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the activity of paclitaxel when administered on a weekly schedule to patients with advanced ovarian cancer who have failed paclitaxel on a 3 or 24 hour infusion schedule. II. Evaluate the toxic effects of paclitaxel when administered on a weekly schedule in this patient population. III. Correlate response with quality of life outcomes, including symptom distress, performance status, and global quality of life.

OUTLINE: This is a single center, open label study. Paclitaxel is administered intravenously every week as a 1 hour infusion. Patients receive prophylactic anti-allergy premedication prior to paclitaxel.

PROJECTED ACCRUAL: 25-30 patients accrued per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or progressive epithelial ovarian cancer defined as: A serial rise in CA 125 over a minimum of 3 samples to a level greater than 50% of the upper limit of normal OR Measurable or evaluable disease Disease progression following paclitaxel given by 3 or 24 hour infusion within the past 6 months

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky at least 60% Life expectancy: Not specified Hematopoietic: AGC at least 1500/uL Platelet count at least 100,000/uL Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Other: No active or uncontrolled infections No history of grade 3-4 peripheral neuropathy of any etiology No previously developed severe hypersensitivity reactions to paclitaxel Not pregnant or lactating Patients of childbearing potential must use effective method of contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior platinum based chemotherapy required Complete recovery from the myelosuppressive effects of prior chemotherapy for a minimum of 3 weeks At least one prior regimen of paclitaxel by 3 or 24 hour infusion within 6 months prior to study, with no intervening chemotherapy Endocrine therapy: No hormone therapy within 3 weeks of entry onto protocol Radiotherapy: No prior radiation therapy to major bone marrow ares within 4 weeks of entry onto protocol Surgery: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-01; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Aghajanian, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States